CLINICAL TRIAL: NCT06983340
Title: Exacerbations and Their Outcomes in Egyptian Patients (EXACOS EG Population): Understanding the Burden of Severe Exacerbations of COPD and the Association Between Frequency of Severe Exacerbations and Clinical and Health-care Utilization Outcomes in Less Well-resourced Countries: Sample of Egyptian Patients.
Brief Title: EXACOS EG Population
Acronym: EXACOS EG
Status: Not yet recruiting | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D5980R00101
Record Dates: First submitted 2025-04-23; First posted 2025-05-21 (Actual); Last update posted 2025-07-15 (Actual); Status verified 2025-07

CONDITIONS: Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Chronic obstructive pulmonary disease (COPD) is a common, progressive disease characterized by airflow obstruction which is not fully reversible. Acute exacerbations of COPD (AECOPD) are described as worsening of COPD symptoms (breathlessness, cough, and sputum volume and purulence) beyond normal day to day variation. Between 30-50% of patients with COPD experience at least one AECOPD per year (1). Even a single moderate AECOPD increases risk of future multiple AECOPD events, starting a spiral of excessive disease progression and leading to an increased risk of death (2). AECOPDs have also been associated with other clinical outcomes such as accelerated lung function decline.

Studies have shown that AECOPDs are related to future AECOPDs, however, little is known about clinical burden and health care utilization in the COPD population. To date, most of published literature reports a combined category of moderate-severe exacerbations, typically stratifying patients as experiencing frequent (i.e., two or more events per patient-year) vs. infrequent (none or one) exacerbations.

In Egypt, COPD is considered one of the most burdensome chronic diseases, with acute exacerbations being directly associated with its burden on patients 'lives. Although no official epidemiological data is available for COPD, its prevalence in Egypt was estimated to be 3.5% in the international epidemiological survey study BREATHE in 2012, while its prevalence in high-risk Egyptian population -defined as population engaged in construction, exposed to biomass fuel, or with smoking history - is estimated to be 9.6%. Moreover, a study reporting on the burden of COPD indicated that the age standardized prevalence of COPD increased by 62% over 3 decades. Regarding AECOPD, studies have explored its reported etiologies and clinical outcomes in Egypt; however, data specifying its incidence and frequency in Egypt is still limited.

ELIGIBILITY:
Inclusion Criteria:

1. are over the age of 40 years old;
2. have had an investigator-confirmed diagnosis of COPD of at least 3 years prior to the index date;
3. have COPD-related data recorded in medical records for at least 3 years prior to the index date, including spirometry (at least one FEV1 measurement) and medication data;
4. have signed a written Informed Consent Form

Exclusion Criteria:

1. have a diagnosis of bronchiectasis, sarcoidosis, Interstitial Lung Diseases, or Idiopathic pulmonary fibrosis. This is because differentiating deteriorations in symptoms/exacerbations in these individuals at attributing them to COPD is impossible.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients, treated by pulmonologists, with an investigator-confirmed diagnosis of COPD for at least 3 years from the index date (the date that signed Informed Consent was obtained) and who meet all of the inclusion and none of the exclusion criteria detailed below will be included. The intention is to study a broad COPD patient population, so minimal eligibility criteria will be applied.
Sampling Method: Non-Probability Sample
Enrollment: 240 (Estimated)
Dates: Start 2025-08-30 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
To estimate the frequency of severe AECOPD in COPD population in Egypt | 3 Years
  The average annual frequency of severe AECOPD will be estimated in the 3 years prior to index date and divided by 3.
To describe any time trends in the frequency of severe exacerbations throughout the 3 years prior to index date | 3 Years
  This will guide the categorization of patients into mutually-exclusive groups of severe AECOPD frequency. We expect the following categories which will be refined upon data descriptive analyses:
  * 0 events
  * 1 severe event
  * 2 severe events
  * 3 severe events
  * >3 severe events The distribution of exacerbations across the entire 3-year period will also be described.

SECONDARY OUTCOMES:
To measure the Modified Medical Research Council (mMRC) dyspnea scale score at time of the study visit | 12 Months
  Medical Research Council (MRC) dyspnea scale grade, as measured during the index date visit
To describe the clinical impact of COPD on the patient | 3 Years
  CAT score as measured during the index date visit
To quantify health care resource utilization by number of severe AECOPD over the 3 years prior to index date. | 3 Years
  • number of emergency department visits
To quantify health care resource utilization by number of severe AECOPD over the 3 years prior to index date. | 3 Years
  • number and length of hospitalizations
To quantify health care resource utilization by number of severe AECOPD over the 3 years prior to index date. | 3 years
  • COPD maintenance prescriptions over the 3 years prior to the index date